CLINICAL TRIAL: NCT03711448
Title: Ustekinumab for the Treatment of Relapse of Refractory Giant Cell Arteritis
Acronym: ULTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAMSON PHRC I 2017
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Patients Relapsing Refractory Giant Cell Arteritis
MeSH Terms: interventions — Prednisone; Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Drug: prednisone treatment; Other: questionnaires; Biological: Blood samples
- Experimental group (Experimental)
  Interventions: Drug: prednisone and ustekinumab treatment; Other: questionnaires; Biological: Blood samples

INTERVENTIONS:
Drug: prednisone treatment — tapering prednisone regimen
  Arms: Control group
Drug: prednisone and ustekinumab treatment — Treatment with prednisone and ustekinumab (90 mg subcutaneously at inclusion (W0), W4, W16 and W28)
  Arms: Experimental group
Other: questionnaires — HAQ ; SF-36 ; FACIT-fatigue
Biological: Blood samples — Additional blood samples for immunomonitoring

SUMMARY:
Giant cell arteritis (GCA) is the most common form of vasculitis after age 50. It is a vasculitis affecting the large vessels, in particular the aorta and its collateral vessels, especially those in the external carotid area.

Corticosteroids are the cornerstone of GCA treatment. They are very effective but are generally continued for 18 to 24 months or more since at least 30% of patients with GCA will relapse during their follow-up. Thus, the vast majority of patients treated for GCA have at least one adverse event from corticosteroid therapy, which is the main source of morbidity in these elderly patients.

Reducing the use of corticosteroids, especially during relapses, is therefore a major objective to improve the treatment of patients with GCA. Methotrexate, abatacept and tocilizumab have been shown to be effective during GCA. However, the therapeutic effect of the first two is modest. As for tocilizumab, its use has many limitations: suspensive effect, many contraindications and there are no biological parameters available for reliable monitoring of inflammatory syndrome in these patients.

Recent data have shown the major role of T helper (Th) Th1 and Th17 T cells in the pathophysiology of GCA. Th17 lymphocytes are sensitive to corticosteroid therapy but Th1 persists despite treatment and produces interferon-γ which activates macrophages and smooth muscle cells, leading to remodelling of the vascular wall responsible for ischemic GCA manifestations. Joint targeting of Th17 and Th1 responses is therefore necessary to fully treat the vascular inflammation that exists during GCA. Ustekinumab, which is a monoclonal antibody blocking the subunit common to IL-12 and IL-23 (p40), blocks the Th1 and Th17 responses, and could therefore be an excellent treatment for GCA.

This study aims to evaluate the efficacy of ustekinumab for the treatment of GCA relapses.

Very little data is available on the use of ustekinumab during GCA. Recently, 14 patients with refractory GCA, defined as the occurrence of at least 2 relapses and the inability to reduce the prednisone dose below 10 mg/d, received ustekinumab treatment. No patients relapsed during treatment while the median dose of prednisone was reduced from 20 to 5 mg/d.

Ustekinumab has also been used successfully in a patient with refractory GCA. Under treatment, the patient did not have a new relapse and the dose of prednisone was reduced. In addition, there was a major decrease in the percentages of circulating Th1 and Th17 lymphocytes.

However, to date, no controlled studies have been conducted to confirm the efficacy of ustekinumab during GCA relapses.

This guarantees the originality and innovation of this study.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Patient with GCA, defined by the following criteria (collected at the time of diagnosis of GCA):

  * Age ≥ 50 years old
  * AND sedimentation rate VS ≥ 50 mm/h or C-reactive protein CRP ≥ 20 mg/L (optional if the temporal artery biopsy (TAB) is positive)
  * AND clinical signs of GCA or signs of rhisomelic pseudopolyarthritis (RPP)
  * AND positive TAB (granulomatous vasculitis lesions) OR evidence of vasculitis of large vessels (aorta or supra-aortic trunks) by angio-TDM, PET-scanner and/or angio-MRI.
* CRP elevation >10 mg/L on at least one occasion during the 6 weeks prior to inclusion
* Relapse treatment initiated less than 6 weeks ago
* Patient with GCA relapse at a dose of prednisone ≤ 20 mg/d and who has received at least 12 consecutive weeks of corticosteroid therapy since the diagnosis of GCA. Relapse is defined as the reappearance of clinical or radiological sign(s) of GCA after a remission phase of at least 1 month AND despite well followed treatment:

  * headache (> 1 day, not relieved by paracetamol and not identical to headache that the patient may have had in the past and that is not related to GCA)
  * hyperesthesia of the scalp, claudication of the jaws or tongue, anomaly of the temporal artery
  * visual signs related to GCA
  * signs of RPP
  * non-infectious fever of more than one week
  * aggravation, recurrence or appearance of signs of vasculitis of large vessels with angioscanner, angio-MRI or PET scanner
  * any other sign related to the activity of the GCA as determined by the investigator

Exclusion Criteria:

* Person not affiliated to or not benefiting from a health insurance system
* Weight < 40kg or > 100kg (at inclusion)
* Non-compliant patient
* Adult unable to express consent
* Patient with a psychotic state not controlled by treatment
* Person subject to a measure of legal protection (curatorship, guardianship)
* Person subject to judicial control
* Women who have not gone through menopause
* Hypersensitivity to ustekinumab, to any of its excipients or to any other murine or human monoclonal antibody
* Latex hypersensitivity (because the packaging of ustekinumab contains latex, which is only present in syringes)
* Relapse with the presence of obvious ophthalmological signs requiring high-dose corticotherapy (1 mg/kg and/or methylprednisolone bolus)
* Surgery scheduled within 12 months (excluding low-risk surgery: endoscopy, bronchoscopy, hysteroscopy, cystoscopy, biopsy or breast surgery, dental care, dental extractions, eye surgery, outpatient surgery, skin surgery)
* Patient with other autoimmune or auto-inflammatory disease (except RPP, autoimmune thyroiditis, Addison's disease, type 1 diabetes, Biermer's disease and presence of autoantibodies without clinical manifestation)
* Neoplasia < 5 years (excluding in situ cervical cancer and skin carcinomas, excluding melanomas, with healthy margin resections [R0]).
* Patient who has received an organ transplant (apart from a corneal transplant)
* Patient who has received an autograft or hematopoietic marrow allograft
* Unstable or poorly controlled disease, acute or chronic, not related to GCA and considered by the investigator as a contraindication to ustekinumab treatment (examples: recurrent infections, ulcers of the lower limbs poorly controlled, unstable ischemic cardiovascular disease, terminal renal failure, liver failure, heart failure ≥ stage III/IV NYHA, diabetes poorly controlled...).
* Other treatments :

  * Patient who has received at least 3 systemic corticoid cures for a condition other than GCA within the last 6 months (dermocorticoids and inhaled corticoids are allowed)
  * Patient receiving long-term corticosteroid treatment (excluding dermocorticoids and inhaled corticosteroids) for a condition other than GCA
  * Patient currently treated or having received, within 4 weeks, cytotoxic, immunosuppressive (except methotrexate and azathioprine which should however be stopped before inclusion), immunomodulatory (except dapsone which should however be stopped before inclusion) or biotherapic treatment.
  * Live vaccine injected within 30 days of inclusion

Infections :

* Chronic (or acute) viral hepatitis B or C
* HIV infection
* Persistent infection or severe infection requiring hospitalization or intravenous antibiotic treatment within 30 days of inclusion (trial antibiotics, regardless of duration and route of administration, are not an exclusion criterion).
* Infection requiring oral antibiotic treatment within 14 days of inclusion (trial antibiotics, regardless of duration and route of administration, are not an exclusion criterion).
* History of histoplasmosis or listeriosis
* Active tuberculosis
* Sign of latent tuberculosis (based on a history of untreated contagion, an opacity greater than 1 cm in diameter on chest X-ray, or a positive in vitro test [QuantiferonR or T-spot-TBR]). A history of tuberculosis disease or latent tuberculosis whose treatment has been completed and which has been properly conducted does not constitute an exclusion criterion, regardless of the outcome of the QuantiferonR or T-spot-TBR.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Percentage of living patients who went into remission after inclusion, without a new relapse and without deviation from the prednisone tapering protocol planned in the study. | Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No